CLINICAL TRIAL: NCT05043987
Title: A Phase 1, Multicenter, Dose Escalation and Dose Expansion Study to Evaluate Safety of CPO102, an Anti-claudin 18.2 Antibody-MMAE Drug Conjugate Administered Intravenously in Patients With Advanced Pancreatic and Gastric Cancers
Brief Title: Dose Escalation and Expansion Study of CPO102, an Anti-claudin 18.2 ADC in Patients With Advanced Cancers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: New IND sponsor to initiate a separate study
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Collaborators: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPO102-US-1001
Record Dates: First submitted 2021-08-30; First posted 2021-09-14 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Cancer; Gastric Cancer
Keywords: Claudin 18.2 ADC; Phase 1; CPO102; Pancreatic Cancer; Gastric Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): Part A will follow the standard 3+3 dose-escalation design and will be enrolled at dose levels of CPO102 at (0.5, 1, 1.8, 2.5, 3.5, 4.5, 5.5 mg/kg).
  Each subject group will receive one dose of CPO-102 every 3 weeks (1 cycle=21 days=1 treatment). For each cohort, the decision whether to dose-escalate will be made once all patients have been enrolled into the cohort and the last patient enrolled has been followed for 21 days (3-week DLT observation period).
  Interventions: Drug: CPO102
- Part B-Arm 1 (Experimental): Upon attaining a RP2D, Part B-Arm 1 will include approximately 15 patients with pancreatic cancer patients. This subject group will receive multiple cycles of a weekly dose of CPO-102 (1 cycle=21 days=1 treatment).
  Interventions: Drug: CPO102
- Part B-Arm 2 (Experimental): Upon attaining a RP2D, Part B-Arm 2 will include approximately 15 gastric (including gastric esophageal junction) cancer patients. This subject group will receive multiple cycles of a weekly dose of CPO-102 (1 cycle=21 days=1 treatment).
  Interventions: Drug: CPO102

INTERVENTIONS:
Drug: CPO102 — Anti-claudin 18.2 Antibody-MMAE Drug Conjugate

SUMMARY:
This Phase 1 study will be a multicenter, single agent, dose escalation and dose expansion study conducted in patients with advanced late stage cancer (pancreatic or gastric including esophageal junction cancers) for which the investigator determines there to be no other standard of care or higher priority therapies available.

DETAILED DESCRIPTION:
This Phase 1 study will be a multicenter, single agent, dose escalation and dose expansion study conducted in patients with advanced late stage cancer (pancreatic or gastric including esophageal junction cancers) for which the investigator determines there to be no other standard of care or higher priority therapies available. All patients must have failed standard first or later lines of systemic therapy.

The study design overview is presented below. The study will consist of 2 parts, Part A and Part B. Part A will explore once every 3 weeks (Q3W) dosing per standard 3+3 dose escalation design. Upon attaining a RP2D, Part B will commence in 2 groups, in approximately 15 patients with advanced pancreatic cancer and 15 patients with advanced gastric including gastric esophageal junction cancers. Part B will seek to confirm the RP2D and will also seek early signals of efficacy in the selected cancer patient populations.

ELIGIBILITY:
Inclusion Criteria:

Applicable to all patients in both Part A and Part B of the study:

* Pathological diagnosis (histological) of pancreatic or gastric including esophageal junction cancers.
* Patient must provide archived tissue block or formalin-fixed paraffin-embedded (FFPE) slides or fresh biopsy prior to start of treatment.
* Positive claudin 18.2 tumor expression defined as ≥50% of tumor cells demonstrating moderate-to-strong membranous staining (2+/3+) by IHC assay performed on sections of tumor derived from formalin fixed paraffin block.
* Adequate organ function.
* Life expectancy >12 weeks.
* Age ≥18 years.
* ECOG performance status 0 or 1 at screening.
* Ability to understand the nature of this study, comply with protocol requirements, and give written informed consent.
* Patients of reproductive potential: All female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before study entry.

Specific criteria for Part A:

* Disease progression or relapse following conventional chemotherapy:

  1. Pancreatic cancer
  2. Gastric cancer (including GEJ cancer)

Specific criteria for Part B:

* Measurable disease suitable for imaging and efficacy tracking as defined by RECIST 1.1
* Disease progression or relapse following conventional chemotherapy:

  1. Pancreatic cancer
  2. Gastric cancer (including GEJ cancer)

Exclusion Criteria:

1. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to baseline or to common terminology criteria for adverse events (CTCAE) grade ≤1, with the exception of alopecia, ≥grade 2 neuropathy, or to the levels dictated in the inclusion/exclusion criteria.
2. Patient has participated in any investigational research study and is being screened for participation within a period of 5 half-lives or 4 weeks, whichever is longer, of the last dose of the investigational therapy.
3. History of severe infusion reaction with monoclonal antibody treatment.
4. Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening), or any uncontrolled infection at screening.
5. HIV positive test within 8 weeks of screening.
6. Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
7. Presence of other active cancers, or history of treatment for invasive cancer ≤3 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (ie, noninvasive) are eligible, as are patients with history of nonmelanoma skin cancer.
8. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
9. Active central nervous system (CNS) disease involvement, defined by cerebrospinal fluid (CSF) cytology, magnetic resonance imaging (MRI) or computerized tomography (CT); patients with asymptomatic CNS metastases are eligible if participants have been clinically stable for at least 4 weeks prior to the first dose of study drug and do not require interventions such as surgery, radiation or any corticosteroid therapy for management of symptoms related to CNS disease.
10. Peripheral neuropathy Grades ≥ 2.
11. Active ocular surface disease at baseline (based on ophthalmic evaluation).
12. Pregnant or nursing (lactating) women.
13. Patients who received claudin 18.2 targeting agents previously.
14. Patients who have received or will receive coronavirus disease 2019 (COVID-19) vaccine within 72 hours prior to the first dose of study drug.
15. Prior radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) during the DLT evaluation period. | through study completion, an average of 3 year
  DLTs are assessed during the first cycle (21 days) in each cohort to determine maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) including Grade ≥ 3, serious, fatal TEAE by relationship. | through study completion, an average of 3 year
  TEAEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v 5.0.
Number of participants with clinically significant changes in vital signs | through study completion, an average of 3 year
  Number of participants with clinically significant changes in vital signs
Number of participants with clinically significant changes in clinical laboratory tests | through study completion, an average of 3 year
  Number of participants with clinically significant changes in clinical laboratory tests
CPO102 pharmacokinetics: Area under the concentration time curve over the dosing interval. | through study completion, an average of 3 year
  CPO102 pharmacokinetics: Area under the concentration time curve over the dosing interval.
CPO102 pharmacokinetics: Maximum concentration of the drug (Cmax) | through study completion, an average of 3 year
  CPO102 pharmacokinetics: Maximum concentration of the drug (Cmax)
CPO102 pharmacokinetics: Time to maximum concentration (Tmax) | through study completion, an average of 3 year
  CPO102 pharmacokinetics: Time to maximum concentration (Tmax)
CPO102 pharmacokinetics: Elimination half-life (t1/2) | through study completion, an average of 3 year
  CPO102 pharmacokinetics: Elimination half-life (t1/2)
CPO102 pharmacokinetics: Clearance (CL) | through study completion, an average of 3 year
  CPO102 pharmacokinetics: Clearance (CL)
CPO102 Objective response rate (ORR) | through study completion, an average of 3 year
  ORR is defined as the proportion of patients in whom a complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 is observed as best overall response.
CPO102 immunogenicity: Number of participants with anti-drug-antibody (ADA) | through study completion, an average of 3 year
  CPO102 immunogenicity: Number of participants with anti-drug-antibody (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Jiangfeng Su, MD, PhD, Study Director — Conjupro Biotherapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No
Undecided